CLINICAL TRIAL: NCT02572505
Title: Pre-Exposure Prophylaxis and Timed Intercourse for HIV-Discordant Couples
Acronym: PrEP-HIVD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Erma Drobnis, Assistant Professional Practice Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #2002937
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: HIV; Infertility
Keywords: HIV-Discordant; Preexposure Prophylaxis
MeSH Terms: conditions — Infertility | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV-Discordant Couple (Experimental): A couple in which the man is HIV-seropositive and the woman is HIV-seronegative who wish to have a biologically related child. Couple will use condoms for all sexual acts except one act of unprotected intercourse during the fertile period when the woman will be taking the drug Truvada.
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Female patient will take Truvada and use condoms for each act of intercourse except once at the optimal time for fertility.
  Other Names: HIV-D; PrEP; Gilead Sciences; emtricitabine; tenofovir disoproxil fumarate

SUMMARY:
Human immunodeficiency virus (HIV) infection has now become a treatable disease and many infected individuals are interested in having a family. Couples in which the man is infected but the woman is HIV-negative (hereafter referred to as HIV-discordant) require medical intervention during procreation to prevent HIV transmission to the female and her child. The current view is that reducing the number of infections involving unprotected intercourse in HIV-discordant couples is a public health issue in the U.S. The safest methods for HIV-discordant couples are insemination using a sperm donor, adoption and remaining childless. However, some couples strongly desire a biologically related child. Fertility clinics in the United States have been resistant to treating HIV-discordant couples, offering only expensive, invasive techniques. This reduces access to care, leading to couples choosing unprotected intercourse to conceive a child. Pre-exposure prophylaxis (PrEP) is a treatment taken by the woman before having unprotected intercourse with an infected man. Truvada has been approved by the Food and Drug Administration (FDA) to reduce the risk of HIV-discordant couples and the Centers for Disease Control and prevention (CDC) has recommended that serodiscordant patients who wish to have a child be counseled on the availability of PrEP. When risks of transmission are minimized, including undetectable HIV in blood and use of PrEP, unprotected intercourse during the fertile period is likely to be a safe option for conceiving a child. The investigators propose to enroll HIV-discordant couples who have been counseled on the safer alternatives of donor insemination, adoption and remaining childless; have been offered referral to a clinic offering sperm washing with insemination or in vitro fertilization (IVF); have been apprised of the risks of using PrEP and one timed intercourse per cycle; and decide to proceed with this method. Couples will be from the population of HIV-discordant patients with a minimal risk of disease transmission as described above. After evaluation for normal fertility and low potential for disease transmission, the couple will receive instruction on timing of the most fertile day of the cycle, and the woman will be given a prescription for the PrEP medication. The woman and any offspring will be followed for 6 months using blood tests to check for evidence of HIV infection.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) infection has now become a treatable disease and many infected individuals are interested in having a family. Couples in which the man is infected but the woman is HIV-negative (hereafter referred to as HIV-discordant) require medical intervention during procreation to prevent HIV transmission to the female and her child. The current view is that reducing the number of infections involving unprotected intercourse in HIV-discordant couples is a public health issue in the U.S.

The risk of HIV transmission by regular intercourse in HIV-discordant couples in a stable relationship is about 1 case for every 1000 sexual acts. However, the risk is extremely low if 1) the couple is monogamous; 2) there is no intravenous (IV) drug use; 3) the man has low HIV viral load, a high CD4 count (CD4 cells are white blood cells that are attacked by HIV), and no symptoms of the disease; 4) the couple is free of other sexually transmitted infections; 5) the male and female genital tracts are free of sores; 6) the man is circumcised; and 7) the man is taking antiretroviral treatment (ART). In fact, studies in African HIV-discordant couples have found no transmission of HIV if patients either have low blood levels of HIV, no symptoms of HIV infection or are taking ART.

The safest methods for HIV-discordant couples are insemination using a sperm donor, adoption and remaining childless. However, some couples strongly desire a biologically related child. Fertility clinics in the U.S. have been resistant to treating HIV-discordant couples. Generally, the available treatment in the U.S. involves in vitro fertilization (IVF), which involves collecting sperm and eggs from the couple and allowing fertilization to occur in the laboratory, with intracytoplasmic sperm injection (ICSI), in which a single sperm is injected directly into the egg. One cycle of treatment costs more than 20% of the median annual income in the U.S., and the birth rate with this method is approximately 35% per cycle of treatment. These factors significantly reduce access to care, and studies have shown that when access to care is low, many couples will choose to use unprotected intercourse, even if counseled on the risks involved. Without appropriate screening and counseling, unprotected intercourse is risky, with 4% of women becoming infected in one study

Pre-exposure prophylaxis (PrEP) is a treatment taken by the woman before having unprotected intercourse with an infected man. The U.S. Food and Drug Administration (FDA) has approved the drug Truvada (Tenofovir/emtricitabine) for use by HIV-discordant couples. Whereas IVF and ICSI are invasive techniques that breach the natural barriers to infection in the female reproductive tract, intercourse preserves these protective mechanisms. The goals of treating HIV-discordant couples are to reduce the infectivity of the male and the susceptibility of the female to infection. Trials carried out primarily in Africa looking at HIV transmission in HIV-discordant couples have shown that use of PrEP significantly reduces the risk of transmission. Based on these results, the U.S. Centers for Disease Control and prevention (CDC) has recommended that serodiscordant patients who wish to have a child be counseled on the availability of PrEP. When risks of transmission are minimized, including undetectable HIV in blood and the use of PrEP, unprotected intercourse during the fertile period is likely to be a safe option for conceiving a child.

An ongoing Swiss trial, started in 2004, has had no infection of the female in 53 couples, and has had an overall pregnancy rate of 75% after 6 cycles of treatment. Preliminary data from a United Kingdom trial reports 13 couples with 11 pregnancies and no female infection. An Italian trial has been initiated recently. Treatment of HIV-discordant couples with PrEP and timed, unprotected intercourse remains experimental.

The investigators propose to enroll HIV-discordant couples who have been counseled on the safer alternatives of donor insemination, adoption and remaining childless; have been offered referral to a clinic offering sperm washing with insemination or ICSI; have been apprised of the risks of using PrEP and one timed intercourse per cycle; and decide to proceed with this method. Couples will be from the population of HIV-discordant patients with a minimal risk of disease transmission as described above. After evaluation for normal fertility and low potential for disease transmission, the couple will receive instruction on timing of the most fertile day of the cycle, and the woman will be given a prescription for the PrEP medication. The woman and any offspring will be followed for 6 months using blood tests to check for evidence of HIV infection.

ELIGIBILITY:
Inclusion Criteria:

Woman:

* 18-40 years of age
* not pregnant
* BMI 18.5-30
* nonsmoker
* no use of IV drugs
* seronegative for HIV
* negative tests for hepatitis C and hepatitis B, human T-lymphotropic virus (HTLV I&II), syphilis, Chlamydia trachomatis and Neisseria gonorrhea
* normal fertility examination
* normal PAP smear and HPV screen

Man:

* 18-50 years of age
* nonsmoker
* no use of IV drugs
* HIV-seropositive
* under the care of an infectious disease specialist
* without evidence of acquired immunodeficiency syndrome (AIDS)
* HIV viral load <50,000 copies/mL and CD4 count > 250 cells/mL for the preceding 6 month period
* taking anti-retroviral medication
* must be circumcised
* have 2 normal semen analyses

Couple:

* must be informed of safer choices (donor insemination, adoption, remaining childless)
* must attest to safe sexual practices.

Exclusion Criteria:

* either man or woman is incarcerated
* either man or woman is unable to provide informed consent
* woman is unable to take Truvada (tenofovir/emtricitabine) medication due to contraindications or adverse reaction

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Proportion of women remaining HIV-seronegative for 6 months after a treatment menstrual cycle | 6 months after each menstrual cycle in which HIV-discordant couple has one act of unprotected intercourse
  After having one act of unprotected intercourse at the woman's fertile period, she will be tested at 6 months by HIV Ab test. Outcome will be reported as proportion of women becoming HIV-seropositive after one cycle of treatment. It is expected that this will be zero.

SECONDARY OUTCOMES:
Proportion of couples achieving pregnancy after each treatment menstrual cycle. | Approximately one month after unprotected intercourse
  If the woman does not start menses after treatment cycle, pregnancy will be measured by serum hCG.

CONTACTS AND LOCATIONS:
Overall Officials: Danny J Schust, M.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- Missouri Center for Reproductive Medicine & Fertility, Columbia, Missouri, United States

REFERENCES:
- [Background] ACOG Committee Opinion no 595: Committee on Gynecologic Practice: Preexposure prophylaxis for the prevention of human immunodeficiency virus. Obstet Gynecol. 2014 May;123(5):1133-1136. doi: 10.1097/01.AOG.0000446855.78026.21. PMID 24785877
- [Background] Practice Committee of American Society for Reproductive Medicine. Recommendations for reducing the risk of viral transmission during fertility treatment with the use of autologous gametes: a committee opinion. Fertil Steril. 2013 Feb;99(2):340-6. doi: 10.1016/j.fertnstert.2012.08.028. Epub 2012 Sep 10. PMID 22975112
- [Background] Barreiro P, Castilla JA, Labarga P, Soriano V. Is natural conception a valid option for HIV-serodiscordant couples? Hum Reprod. 2007 Sep;22(9):2353-8. doi: 10.1093/humrep/dem226. Epub 2007 Jul 19. PMID 17640945
- [Background] Daar ES, Daar JF. Human immunodeficiency virus and fertility care: embarking on a path of knowledge and access. Fertil Steril. 2006 Feb;85(2):298-300; discussion 301. doi: 10.1016/j.fertnstert.2005.08.018. PMID 16595202
- [Background] De Carli G, Palummieri A, Liuzzi G, Puro V. Safe conception for human immunodeficiency virus-discordant couples: the preexposure prophylaxis for conception alternative. Am J Obstet Gynecol. 2014 Jan;210(1):90. doi: 10.1016/j.ajog.2013.08.011. Epub 2013 Aug 14. No abstract available. PMID 23954529
- [Background] de Vincenzi I. A longitudinal study of human immunodeficiency virus transmission by heterosexual partners. European Study Group on Heterosexual Transmission of HIV. N Engl J Med. 1994 Aug 11;331(6):341-6. doi: 10.1056/NEJM199408113310601. PMID 8028613
- [Background] Del Romero J, Castilla J, Hernando V, Rodriguez C, Garcia S. Combined antiretroviral treatment and heterosexual transmission of HIV-1: cross sectional and prospective cohort study. BMJ. 2010 May 14;340:c2205. doi: 10.1136/bmj.c2205. PMID 20472675
- [Background] Downs AM, De Vincenzi I. Probability of heterosexual transmission of HIV: relationship to the number of unprotected sexual contacts. European Study Group in Heterosexual Transmission of HIV. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Apr 1;11(4):388-95. doi: 10.1097/00042560-199604010-00010. PMID 8601226
- [Background] Frodsham LC, Boag F, Barton S, Gilling-Smith C. Human immunodeficiency virus infection and fertility care in the United Kingdom: demand and supply. Fertil Steril. 2006 Feb;85(2):285-9. doi: 10.1016/j.fertnstert.2005.07.1326. PMID 16595198
- [Background] Gilling-Smith C, Nicopoullos JD, Semprini AE, Frodsham LC. HIV and reproductive care--a review of current practice. BJOG. 2006 Aug;113(8):869-78. doi: 10.1111/j.1471-0528.2006.00960.x. Epub 2006 Jun 2. PMID 16753050
- [Background] Gray RH, Wawer MJ, Brookmeyer R, Sewankambo NK, Serwadda D, Wabwire-Mangen F, Lutalo T, Li X, vanCott T, Quinn TC; Rakai Project Team. Probability of HIV-1 transmission per coital act in monogamous, heterosexual, HIV-1-discordant couples in Rakai, Uganda. Lancet. 2001 Apr 14;357(9263):1149-53. doi: 10.1016/S0140-6736(00)04331-2. PMID 11323041
- [Background] Klein J, Pena JE, Thornton MH, Sauer MV. Understanding the motivations, concerns, and desires of human immunodeficiency virus 1-serodiscordant couples wishing to have children through assisted reproduction. Obstet Gynecol. 2003 May;101(5 Pt 1):987-94. doi: 10.1016/s0029-7844(03)00012-7. PMID 12738162
- [Background] Lampe MA, Smith DK, Anderson GJ, Edwards AE, Nesheim SR. Achieving safe conception in HIV-discordant couples: the potential role of oral preexposure prophylaxis (PrEP) in the United States. Am J Obstet Gynecol. 2011 Jun;204(6):488.e1-8. doi: 10.1016/j.ajog.2011.02.026. Epub 2011 Mar 31. PMID 21457911
- [Background] Mandelbrot L, Heard I, Henrion-Geant E, Henrion R. Natural conception in HIV-negative women with HIV-infected partners. Lancet. 1997 Mar 22;349(9055):850-1. doi: 10.1016/S0140-6736(05)61754-0. No abstract available. PMID 9121267
- [Background] Mastro TD, de Vincenzi I. Probabilities of sexual HIV-1 transmission. AIDS. 1996;10 Suppl A:S75-82. doi: 10.1097/00002030-199601001-00011. No abstract available. PMID 8883613
- [Background] Quinn TC, Wawer MJ, Sewankambo N, Serwadda D, Li C, Wabwire-Mangen F, Meehan MO, Lutalo T, Gray RH. Viral load and heterosexual transmission of human immunodeficiency virus type 1. Rakai Project Study Group. N Engl J Med. 2000 Mar 30;342(13):921-9. doi: 10.1056/NEJM200003303421303. PMID 10738050
- [Background] Royce RA, Sena A, Cates W Jr, Cohen MS. Sexual transmission of HIV. N Engl J Med. 1997 Apr 10;336(15):1072-8. doi: 10.1056/NEJM199704103361507. No abstract available. PMID 9091805
- [Background] Saracco A, Veglia F, Lazzarin A. Risk of HIV-1 transmission in heterosexual stable and random couples. The Italian Partner Study. J Biol Regul Homeost Agents. 1997 Jan-Jun;11(1-2):3-6. No abstract available. PMID 9418153
- [Background] Sauer MV. Sperm washing techniques address the fertility needs of HIV-seropositive men: a clinical review. Reprod Biomed Online. 2005 Jan;10(1):135-40. doi: 10.1016/s1472-6483(10)60815-2. PMID 15705311
- [Background] Vernazza PL, Hollander L, Semprini AE, Anderson DJ, Duerr A. HIV-discordant couples and parenthood: how are we dealing with the risk of transmission? AIDS. 2006 Feb 28;20(4):635-6. doi: 10.1097/01.aids.0000210625.06202.c2. No abstract available. PMID 16470136
- [Background] Vernazza PL, Graf I, Sonnenberg-Schwan U, Geit M, Meurer A. Preexposure prophylaxis and timed intercourse for HIV-discordant couples willing to conceive a child. AIDS. 2011 Oct 23;25(16):2005-8. doi: 10.1097/QAD.0b013e32834a36d0. PMID 21716070
- [Background] Wawer MJ, Gray RH, Sewankambo NK, Serwadda D, Li X, Laeyendecker O, Kiwanuka N, Kigozi G, Kiddugavu M, Lutalo T, Nalugoda F, Wabwire-Mangen F, Meehan MP, Quinn TC. Rates of HIV-1 transmission per coital act, by stage of HIV-1 infection, in Rakai, Uganda. J Infect Dis. 2005 May 1;191(9):1403-9. doi: 10.1086/429411. Epub 2005 Mar 30. PMID 15809897
- [Background] Whetham J, Taylor S, Charlwood L, Keith T, Howell R, McInnes C, Payne E, Home J, White D, Gilleece Y. Pre-exposure prophylaxis for conception (PrEP-C) as a risk reduction strategy in HIV-positive men and HIV-negative women in the UK. AIDS Care. 2014;26(3):332-6. doi: 10.1080/09540121.2013.819406. Epub 2013 Jul 22. PMID 23876052